CLINICAL TRIAL: NCT01295879
Title: Effect of Ergocalciferol Repletion on Urine Calcium Among Stone Formers With Vitamin D Deficiency and Hypercalciuria
Brief Title: Vitamin D Repletion in Stone Formers With Hypercalciuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, David E. Leaf, Nephrology Fellow, New York Presbyterian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF3346
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Nephrolithiasis; Urolithiasis; Idiopathic Hypercalciuria; Vitamin D Deficiency; Disorder of Vitamin D
Keywords: Vitamin D insufficiency
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis; Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ergocalciferol (Experimental): Subjects will take Ergocalciferol (vitamin D), 50,000 IU's orally per week for 8 weeks
  Interventions: Drug: Ergocalciferol

INTERVENTIONS:
Drug: Ergocalciferol — Ergocalciferol 50,000 IU's orally per week, for 8 weeks
  Other Names: Vitamin D2

SUMMARY:
Vitamin D plays a critical role in maintaining bone health, as well as preventing cardiovascular disease, cancer, and various autoimmune diseases, such as diabetes. Vitamin D deficiency is very common in the United States and worldwide, and is now being increasingly recognized and treated. One group in which vitamin D deficiency may be particularly important is patients who have had kidney stones. These patients frequently have elevated levels of calcium in their urine, which is a common and important risk factor for calcium containing kidney stones. Because vitamin D increases absorption of calcium into the blood by the intestines, physicians may be reluctant to prescribe vitamin D therapy to patients with vitamin D deficiency if they also have kidney stones and high amounts of calcium in the urine. They are concerned about the possible risk of increasing the amount of calcium in the urine (and thereby increasing the risk of calcium stones occurring again). However, studies in patients without kidney stones, as well as studies in patients with high calcium levels in the urine, have demonstrated that giving vitamin D is effective and safe and does not increase calcium in the urine. Therefore, the investigators will study the effects of giving vitamin D on the amount of calcium in the urine in patients with a history of kidney stones and elevated calcium in the urine. The investigators will evaluate the safety of giving vitamin D to this particular group of patients.

DETAILED DESCRIPTION:
The investigators plan to conduct a clinic-based interventional study of 30 patients followed at outpatient urology clinics associated with New York Presbyterian Hospital (NYPH). The intervention is supplementation with oral ergocalciferol 50,000 IU per week for 8 weeks, and each participant will serve as his/her own control. The formulation, dose, and duration of vitamin D therapy is reflective of that which is given in routine clinical practice to patients with vitamin D deficiency. The outcome is the change in urinary calcium excretion.

ELIGIBILITY:
Inclusion Criteria:

* History of nephrolithiasis as per medical record
* Urinary calcium excretion between 150 and 400 mg/day (measured within 3 months of study enrollment)
* 25(OH)D deficiency or insufficiency (defined as a serum level < 30 ng/ml) within 3 months of enrollment

Exclusion Criteria:

* Pregnant women, since the optimal dose of vitamin D supplementation in this population has not been rigorously studied.
* Known uric acid, cystine, or struvite stone disease (because our intervention is predominantly aimed at patients with calcium stone disease). An exception to this is patients who have passed both uric acid and calcium stones, or patients who have passed stones of mixed composition (uric acid and calcium).
* Hypercalcemia (serum calcium > 10.4 mg/dL) at baseline
* Acute stone event or gross hematuria (blood in the urine) within the past 2 months
* Recent stone intervention within the past 1 month
* Suspected or known secondary causes of hypercalciuria, such as primary hyperparathyroidism, sarcoidosis, hyperthyroidism, or malignancy (except nonmelanoma skin cancer)
* Addition or dose change of medicines potentially affecting urinary calcium since the baseline 24hour urine collection (including diuretics, magnesium supplements, potassium supplements, potassium citrate, and vitamin D supplementation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ergocalciferol
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ergocalciferol
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in 24 Hour Urine Calcium
Description: Elevated values of urine calcium are a risk factor for recurrence of calcium kidney stones
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Ergocalciferol
Number analyzed (Participants) | 29
mg/day | 2 (71)

2. Secondary Outcome: Change in 24 Hour Urine Supersaturation of Calcium Oxalate
Description: Elevated values of calcium oxalate supersaturation in the urine are a risk factor for recurrence of calcium kidney stones
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: (unitless)
Arm/Group | Ergocalciferol
Number analyzed (Participants) | 29
(unitless) | -1 (3.5)

3. Secondary Outcome: Recurrence of Kidney Stones
Time Frame: 8 weeks
Measure: Number; unit: # of stone recurrences
Arm/Group | Ergocalciferol
Number analyzed (Participants) | 29
# of stone recurrences | 0

ADVERSE EVENTS:
Arm/Group | Ergocalciferol
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes